CLINICAL TRIAL: NCT04394364
Title: Analysis and Record Intraoperative Bispectral Index of Patients of Thoracic Surgeries
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020-02-018AC
Record Dates: First submitted 2020-03-03; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Bispectral Index and Neurmuscular Monitoring Data in Anesthetized Patients
MeSH Terms: interventions — Consciousness Monitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- BIS monitor group: Patients under monitoring of BIS
  Interventions: Device: Bispectral index

INTERVENTIONS:
Device: Bispectral index — The BIS monitor will be attached to patients' forehead before anesthetized and kept until the end of the surgery

SUMMARY:
Bispectral index(BIS) is commonly used to monitor the depth of anesthesia. The electroencephalographic signal is collected and analyzed by the device, resulting a number related to the awareness of the patient. Electromyography is also recorded. The aim of the study is recording and analyzing the data of BIS and try to find it's relation to intraoperative neuromuscular blockade.

ELIGIBILITY:
Inclusion Criteria:

* ASA class between 1 and 3
* Patients scheduled for chest surgery

Exclusion Criteria:

* Neuromuscular diseases
* Mental and psychiatric disturbance
* ASA class over 4
* Drug abuse
* Aboriginals

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing chest surgeries
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Establishing the predicting model of intraoperative electromyographics of BIS monitor and train-of-four of neuromuscular transmission monitor | six months
  We will collect EMG activity of bispectral index and train-of-four/count of neuromuscular trasmission monitor in patients undergoing pulmonary surgeries. Total intravenous anesthesia will be given to all included patients, and data will be collected since the induction of anesthesia until extubation of endotracheal tube.By statistical methods, we expect to establish the model predicting intraoperative neuromuscular blockade by EEG activity of BIS monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared to other researchers